CLINICAL TRIAL: NCT05968820
Title: Tailoring a Sleep Health Enhancement Intervention for Older Adults to Address Frailty
Brief Title: Sleep Health Enhancement in Older Adults to Address Frailty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Catherine Siengsukon, PT, PhD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00150428
Record Dates: First submitted 2023-07-18; First posted 2023-08-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Frailty
Keywords: Sleep Health; Older Adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Health Enhancement Intervention (Experimental): The sleep health enhancement intervention is a 4-week, 1x/week one-one-one program with a graduate research assistant who will be trained and supervised by the PI in provision of the sleep health enhancement intervention.
  Interventions: Behavioral: Sleep Health Enhancement Intervention
- Wait-List Control Group (No Intervention): The wait-list control group will be encouraged to continue with their usual activities and sleep habits during the wait period between baseline and reassessment and will undergo the sleep health enhancement intervention following the initial reassessment.

INTERVENTIONS:
Behavioral: Sleep Health Enhancement Intervention — The program is based on principles from CBT-I (time in bed restriction, stimulus control, relaxation techniques, sleep education) and includes behavioral strategies to entrain circadian rhythm, strengthen sleep homeostasis, reduce hyperarousal, and sleep hygiene techniques. Self-Determination Theory (SDT) and Social Cognitive Theory (SCT) will serve as the theoretic framework for behavior change techniques (BCT) threaded through the sleep health enhancement intervention. Participants will maintain a sleep diary during the program to aid in tailoring the program, self-monitoring of behavior, and feedback of behavior. Goals will be set by the participant at each session and reviewed at subsequent sessions, and motivational interviewing principles will be incorporated.
  Arms: Sleep Health Enhancement Intervention

SUMMARY:
The objective of the proposed study is to tailor a sleep health enhancement intervention to older adults and assess preliminary efficacy on reducing frailty in older adults. This pilot study will be conducted in two stages. In the treatment development stage, we will recruit n=10 older individuals age ≥65 with poor sleep health (≤ 7 on the Ru-SATED self-report questionnaire) to assess acceptability and tailor the sleep health enhancement intervention for older adults. In the pilot study stage to assess preliminary efficacy of the tailored sleep health enhancement intervention, n=30 older adults with poor sleep health will be randomly assigned to a 4-week 1x/week, telehealth-delivered sleep health enhancement intervention or to a wait-list control condition. Participants will wear wrist-worn actigraphy, complete sleep, frailty, and quality of life questionnaires at baseline and reassessments.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* ≤ 7 on the RU-SATED self-report questionnaire
* MMSE ≥25 and AD8 <3

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea or restless leg syndrome)
* >3 on the STOP BANG indicating increased risk of sleep apnea
* Evidence of restless legs syndrome on RLS-Diagnosis Index
* Evidence of circadian rhythm sleep-wake disorder
* Evidence of parasomnia
* Regular use (>2x/week) of prescription or over-the-counter medications to improve sleep
* Score of ≥15 on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorse any suicidal ideation (answer 1, 2 or 3 on #9 of the PHQ-9)
* Score of ≥10 on the Generalized Anxiety Disorder (GAD-7) indicating moderate to severe anxiety
* Self-report of current or history (up to 2 years) of drug or alcohol abuse based on the DSM-V criteria
* History of nervous system disorder such as stroke or Parkinson's disease
* Severe mental illness such as schizophrenia or bipolar disorder
* Current or history (within 5 years) of shift work including hours of midnight-4am
* Is currently receiving a behavioral sleep health intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
6-item Acceptability Scale | 6 week
  5-point Likert scale on ease of use, understandability, enjoyment, perceived helpfulness, time commitment, and overall satisfaction
semi-standardized qualitative interview | 6 week
  Feasibility and acceptability will be assessed via semi-structured interview with a trained graduate research assistant following standard qualitative methods to determine attitudes, perceptions and experiences of effectiveness, potential barriers, benefits, and likes/dislikes of the sleep health enhancement intervention. The interview will be recorded for analysis purposes
Tilburg Frailty Indicator | baseline, 6 week and 12 week reassessments
  The Tilburg Frailty Indicator consists of 15 questions with score ranging from 0-15 with a higher score indicating higher level of frailty. The physical, psychological, and social frailty sub scores range from 0-8, 0-4, and 0-3 respectively.
WHOQOL-BREF | baseline, 6 week and 12 week reassessments
  The WHOQOL-BREF consists of 26 items and 4 domains of quality of life (psychological, physical health, social relationships and environmental). Scores range from 4-20 for each domain and a higher score indicates higher quality of life.
Ru_SATED sleep health composite | baseline, 6 week and 12 week reassessments
  Ru-SATED sleep health composite will be calculated using actigraphy data and self-report questionnaires. The domains will be summed to create the composite sleep health score ranging from 0-6 with a higher score indicating better sleep health.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | baseline, 6 week and 12 week reassessments
  Scores range from 0-21 with a higher score indicating a lower quality of sleep. A global score of >5 indicates poor sleep quality.
Epworth Sleepiness Scale | baseline, 6 week and 12 week reassessments
  Consists of eight scenarios of daily activity, and participants use a four-point Likert scale to rate how likely they are to doze. Score ranges 0-24 with a higher score indicating daytime sleepiness.
Dysfunctional Beliefs About Sleep | baseline, 6 week and 12 week reassessments
  This assessment is a 10 item Likert-scale self-report questionnaire. Higher scores indicate more dysfunctional beliefs.
Sleep Self-Efficacy | baseline, 6 week and 12 week reassessments
  Sleep Self-Efficacy is a 9 item self-report Likert-scale questionnaire use to identify sleep self-efficacy. Scores range from 0-45 and a higher score indicates higher sleep self-efficacy.
Actigraphy | baseline, 6 week and 12 week reassessments
  Participants will wear an actigraph on their non-dominant wrist for 7 nights

OTHER OUTCOMES:
Timed Up and Go | baseline, 6 week and 12 week reassessments
  Timed Up and Go measures functional mobility and consists of sitting in a chair, standing up, walking 3-m, turning around, returning to the chair, and sitting down. The outcome is the time in seconds it takes to complete the task.
15 ft walk test | baseline, 6 week and 12 week reassessments
  The test is performed in a hallway or open space, and the time it takes to walk 15 ft is noted in seconds.
6-Minute Walk Test (6MWT) | baseline, 6 week and 12 week reassessments
  The test is performed in a hallway or open space with two cones marking the turn-around points. The participant walks between the two cones for six minutes. Distance is measured by number of laps completed.
Grip strength of the dominant and nondominant hand | baseline, 6 week and 12 week reassessments
  Grip strength of the dominant and nondominant hand will be assessed using a dynamometer with the participant seated, elbow flexed to 90 degrees, and arm by their side. The participant will perform one practice submaximal effort for acclimation followed by one maximal effort squeeze.
The Continuous Performance Test (CPT) | baseline, 6 week and 12 week reassessments
  The Continuous Performance Test (CPT) requires participants to respond as quickly and accurately as possible to a series of stimuli that are delivered via computer. The participants will be instructed to tap the space bar for every letter except "X." The participants' scores will be determined by their scores in detectability (e.g., difficulty differentiating targets from non-targets), error type (e.g., omissions, commissions, perseverations) and reaction time statistics.
The Stroop Test | baseline, 6 week and 12 week reassessments
  The Stroop Test requires participants to inhibit the natural response (reading a word) and replace it with another response (saying a color). Each participant is given a list of X's printed in colored ink and a list of words printed in colored ink. The participant is instructed to name the color of the ink. They are given 45 seconds to name as many colors as they can. The reported outcome measure of this test is an interference score that is the difference between the two conditions while normalizing for number of x's using the following formulae: x-words/x.
Cognitive Failures Questionnaire (CFQ) | baseline, 6 week and 12 week reassessments
  Cognitive Failures Questionnaire (CFQ) assesses perception of cognitive abilities over the past 6 months. consists of 25 items that the individual rates on a 5-point Likert scale with 0 = "never" and 4 = "Very Often" with a summary score of 0-100 with a higher score indicating poorer perceived cognitive abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center- Sleep, Health and Wellness Laboratory, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No